CLINICAL TRIAL: NCT05254990
Title: Reparixin 1200 mg TID as add-on to SoC to Limit Disease Progression in Hospitalised Patients With COVID-19 and Other Community-Acquired Pneumonia. A Multicentre, Randomised, Double-blinded, Placebo-controlled, Phase III Trial (REPAVID-22)
Brief Title: Reparixin add-on Therapy to Std Care to Limit Progression in Pts With COVID19 & Other Community Acquired Pneumonia
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was stopped due to futility as per protocol
Sponsor: Dompé Farmaceutici S.p.A (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: REP0321; 2021-006951-32 (EudraCT Number)
Record Dates: First submitted 2022-02-22; First posted 2022-02-24 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Infectious Pneumonia; Severe COVID-19
Keywords: COVID-19; SARS-CoV-2; Infectious pneumonia acquired in the community (CAP)
MeSH Terms: conditions — COVID-19 | interventions — reparixin

STUDY DESIGN:
Intervention Model Description: male and female patients >18 years, hospitalised for COVID-19, will be assigned (1:1) to receive either oral reparixin (treatment group) or matched placebo (control group) three times a day (TID) for up to 21 days.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Reparixin + standard of care (Experimental): Reparixin will be administered orally at the dose of 1200 mg (2 x 600 mg tablets) TID (6 tablets daily) for up to 21 days.
  The three daily doses will be administered maintaining an interval between doses of about 8 hours.
  Interventions: Drug: Reparixin
- Placebo + standard of care (Placebo Comparator): Placebo tablets are identical in appearance to the active formulation. Placebo will be administered with the same treatment schedule.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Reparixin — Reparixin 600 mg tablets, administered orally at the dose of 1200 mg TID (2 tablets TID) as add-on therapy to standard of care up to 21 days. IMP can be taken with a glass of water (about 250 mL) and a light meal or snack, as it is preferable that reparixin is taken with food. However, if the patient is unable to eat, the study drug may still be administered without concomitant food ingestion.
  Other Names: Repertaxin L-lysine salt
  Arms: Reparixin + standard of care
Other: Placebo — Administered orally three times a day (TID) as add-on therapy to standard of care up to 21 days.
  Placebo can be taken with a glass of water (about 250 mL) and a light meal or snack, as it is preferable that placebo is taken with food. However, if the patient is unable to eat, the placebo may still be administered without concomitant food ingestion.
  Other Names: Matched placebo
  Arms: Placebo + standard of care

SUMMARY:
Primary objective:

- To evaluate the efficacy of oral reparixin versus standard care alone in limiting disease progression in adult patients hospitalised for infectious pneumonia acquired in the community (CAP), including COVID-19.

Secondary objectives:

- To determine the effect of reparixin on several disease severity/progression measures including recovery, ventilatory free days and mortality.

Safety objectives:

- To evaluate the safety of oral reparixin versus placebo in the specific clinical setting.

DETAILED DESCRIPTION:
Multinational, multicentre, randomised, double-blind, placebo-controlled, parallel-group, phase III trial.

It will enrol 526 male and female patients >18 years, hospitalised for CAP (including COVID-19), assigned (1:1) to receive either oral reparixin (treatment group) or matched placebo (control group) three times a day (TID) for up to 21 days. Randomisation will be stratified according to disease severity and site.

All the patients will receive the standard of care based on their clinical need, including COVID-19 and CAP medications, as per local standard therapy at the trial site and in line with international guidelines.

The primary outcome will be evaluated at day 28, secondary will be evaluated from day 3 to day 180.

An independent external data monitoring committee (DMC) will oversee the study and evaluate unblinded interim data for efficacy, futility, and safety.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent signed
2. Male and female ≥18 years old;
3. Patients hospitalized for clinically suspected CAP, defined as the occurrence of (within 48h from hospital admission):

   1. at least 1 of the following signs/symptoms: dyspnea, cough, purulent sputum, crackles (rales) and/or rhonchi
   2. body temperature > 38°C or <36°C (before or during admission) or leucocytosis (> local ULN)
   3. new/increased pulmonary infiltrate(s) by chest imaging
4. Need for non-invasive supplemental oxygen (NIAID-OS 5-6; Appendix 14.4.1);
5. SpO2 <92% at room air, or PaO2/FiO2 (or SpO2/FiO2) <300;
6. Females of child-bearing potential and with an active sexual life must not wish to get pregnant within 30 days after the end of the study and must be using at least one of the following reliable methods of contraception:

   1. Hormonal contraception, systemic, implantable, transdermal, or injectable contraceptives for at least 2 months before the screening visit until 30 days after the last IMP dose
   2. A non-hormonal intrauterine device [IUD] or female condom with spermicide or contraceptive sponge with spermicide or diaphragm with spermicide or cervical cap with spermicide for at least 2 months before the screening visit until 30 days after the last IMP dose
   3. A male sexual partner who agrees to use a male condom with spermicide
   4. A sterile sexual partner

Female participants of non-child-bearing potential or in post-menopausal status for at least 1 year will be admitted. For all female subjects, with child-bearing potential, pregnancy test result must be negative before first drug intake.

Exclusion Criteria:

1. Treatment with IMV or ECMO (NIAID-OS 7);
2. Hepatic dysfunction: ALT or AST > 5 ULN; history of chronic hepatic disease (defined with Child-Pugh score B or C);
3. Renal dysfunction: estimated glomerular filtration rate (eGFR, MDRD) <50 mL/min/1.73 m2, or need for haemodialysis or hemofiltration;
4. Current use of >2 immunosuppressive medications or immunosuppression status (AIDS, aplastic anaemia, asplenia, systemic chemotherapy within the past 3 months, neutropenia (ANC < local LLN), solid organ or bone marrow transplant recipients)
5. Treatment with prohibited medication within 5 half-lives, and inability to stop during treatment period (see section 5.5.2);
6. Anticipated discharge from the hospital or transfer to another hospital within 72 hours of screening
7. History of:

   1. intolerance or hypersensitivity to ibuprofen to more than one medication belonging to the class of sulfonamides, such as sulfamethazine, sulfamethoxazole, sulfasalazine, nimesulide or celecoxib (hypersensitivity to sulphanilamide antibiotics alone, e.g. sulfamethoxazole does not qualify for exclusion)
   2. lactase deficiency, galactosemia or glucose-galactose malabsorption
   3. gastrointestinal bleeding or perforation due to previous NSAIDs therapy or recurrent peptic ulcer/haemorrhage
   4. allergy to reparixin or any component of the IMP formulation
8. Active bleeding or bleeding diathesis (excluding menses), prior intracranial haemorrhage
9. Participation in other interventional clinical trials
10. Clinical condition not compatible with oral administration of the study drug
11. Pregnancy:

    1. positive or missing pregnancy test before first drug intake or day 1;
    2. pregnant or lactating women;
    3. women of childbearing potential and fertile men who do not agree to use at least one primary form of contraception for the duration of the study
12. Current hospital stay >72h
13. Complicated CAP-associated conditions, such as fungal pulmonary infection, tuberculosis infection, abscess, empyema, significant bilateral pleural effusion, massive pulmonary embolism

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 409 (Actual)
Dates: Start 2022-04-27 (Actual); Primary Completion 2024-09-27 (Actual); Study Completion 2024-09-27 (Actual)

PRIMARY OUTCOMES:
Proportion of patients dead or requiring Invasive Mechanical Ventilation (IMV) or Extracorporeal Membrane Oxygenation (ECMO) by day 28 [NIAID-OS 7]. | Day 28
  NIAID-OS = National Institute of Allergy and Infectious Disease - Ordinal Scale

SECONDARY OUTCOMES:
All-cause mortality at day 180 | Day 180
Proportion of patients alive and discharged at day 28 | Day 28
Ventilatory-free days (VFD) at day 28 | Day 28
  Number of days from Day 0 to Day 28 when the patient will alive and free of invasive ventilation. In case of multiple periods of IMV during the first 28 days, the total duration of ventilation considered all periods of ventilation during the index admission. Patients who will die within 28 days or will be still on invasive ventilation after 28 days will score zero VFDs18
Occurrence of IMV (or ECMO) by day 28 | Day 28
Length of primary hospital stay | Throughout the trial
Clinical failure by day 3 and day 7 | day 3 and day 7
  Clinical failure will be defined as the occurrence of IMV/ECMO or vasopressor, or death
28-day ICU-free days | Day 28
Days free of IMV/ECMO (number of days with NIAID-OS 1-6) at day 28 | Day 28
Duration of antibiotic therapy (days) at day 28 | Day 28
Hospital free days | Day 28
Proportion of patients recovered | days 3, 7±1, 14±2, 21±2, 28 ±2 or at hospital discharge
  downward shift from screening of ≤2 points on the NIAID-OS or live discharge from hospital)
Proportion of patients worsening | days 3, 7±1, 14±2, 21±2, 28 ±2 or at hospital discharge
  upward shift from screening of at least >1 point of the NIAID-OS)
PO2/FiO2 | days 3, 7±1, 14±2, 21±2, 28 ±2 or at hospital discharge
All-cause mortality | Days 28 and 90
Hospital re-admission by day 90 and 180 | Days 90 and 180
Time to discharge or to a NEWS of ≤ 2 (for 24 hours), whichever occurs first | Day 28
Change in inflammatory markers (LDH, CRP, ferritin; D-dimer, PCT) and cytokines | Days 3, 7±1, 14±2, 21±2, 28±2 or at hospital discharge]
Change in quality of life using EuroQol-5-dimensions-5 levels (EQ-5D-5L) questionnaire | 90±7 and 180±14 days
  The EQ-5D-5L asks patients to indicate whether they have no, slight, moderate, severe, extreme problems on each of five dimensions of health: mobility; self-care; usual activities; pain/discomfort; anxiety/depression.
Duration of IMV and/or ECMO at 90 and 180 days | Days 90 and 180
ICU admission at 90 and 180 days | Days 90 and 180
ICU length of stay at 90 and 180 days | Days 90 and 180
Hospital length of stay at 90 and 180 days | Days 90 and 180
Occurrence of infections at 90 and 180 days | Days 90 and 180

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Landoni, MD, Principal Investigator — IRCCS Ospedale San Raffaele Centro di Ricerca Anestesia e Rianimazione
Locations (101):
- United States (40):
  - MD Banner University Medical Center /Arizona University, Tucson, Arizona
  - UC Davis Medical Center - UC Davis Medical Group - Davis, Davis, California
  - University of Southern California, Los Angeles, California
  - UCI Health, Orange, California
  - Denver Health, Denver, Colorado
  - Nuvance Health, Danbury, Connecticut
  - MedStar Health Research Institute-Hyatteville, Maryland, Washington D.C., District of Columbia
  - Research Alliance Inc., Clearwater, Florida
  - University of Florida-Jacksonville, Jacksonville, Florida
  - University of South Florida, Tampa, Florida
  - Emory Johns Creek Hospital, Atlanta, Georgia
  - Augusta University Health - Augusta University Medical Center, Augusta, Georgia
  - Northwestern University, Feinberg School of Medicine, Chicago, Illinois
  - Jesse Brown VA Medical Center, Chicago, Illinois
  - Insight Hospital & Medical Center Chicago, Chicago, Illinois
  - Northshore University HealthSystem, Evanston, Illinois
  - Methodist Hospital, Gary, Indiana
  - Norton Healthcare, Louisville, Kentucky
  - Tufts Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Newton-Wellesley Hospital, Newton, Massachusetts
  - NorthStar Anesthesia / Detroit Medical Center, Detroit, Michigan
  - MidMichigan Medical Center - Midland, Midland, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - University Hospital - MU Healthcare, Columbia, Missouri
  - Washington University, School of Medicine, St Louis, Missouri
  - Mercy Research St Louis, St Louis, Missouri
  - NYU Langone Hospital-Brooklyn, Brooklyn, New York
  - New York University Langone Health, New York, New York
  - Duke University Hospital, Durham, North Carolina
  - University of Oklahoma Medical Center, Oklahoma City, Oklahoma
  - Oregon Health & Science University (OHSU) - Pulmonary Clinic, Portland, Oregon
  - Jefferson University Hospital, Philadelphia, Pennsylvania
  - University of Tennessee Medical Center, Knoxville, Tennessee
  - Baptist Hospitals of Southeast Texas, Beaumont, Texas
  - Texoma Medical Center, Denison, Texas
  - University of Utah Hospitals & Clinics, Salt Lake City, Utah
  - University of Virginia Medical Center, Charlottesville, Virginia
  - Virginia Commonwealth University Health, Richmond, Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Argentina (18):
  - Hospital Interzonal General de Agudos Dr Jose Penna, Bahía Blanca, Buenos Aires
  - CEMIC, Ciudad Autonoma Buenos Aires, Buenos Aires
  - Hospital Italiano de Buenos Aires, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Hospital Italiano de La Plata, La Plata, Buenos Aires
  - Instituto Medico Platense, La Plata, Buenos Aires
  - Clinica Independencia, Munro, Buenos Aires
  - Sanatorio Finochietto, Ciudad Autonoma de Buenos Aire, Buenos Aires F.D.
  - Hospital Aleman, Buenos Aires, Ciudad Autonoma Buenos Aires
  - Sanatorio de la Cañada, Villa María, Córdoba Province
  - Sanatorio Britanico S.A., Rosario, Santa Fe Province
  - Clinica Mayo de Urgencias Medicas Cruz Blanca SRL, San Miguel de Tucumán, Tucumán Province
  - Clinica Adventista Belgrano, Buenos Aires
  - Sanatorio Agote, Buenos Aires
  - Hospital Britanico de Buenos Aires, Ciudad Autonoma Buenos Aires
  - Clinica Chutro, Córdoba
  - Nuevo Hospital San Roque, Córdoba
  - Sanatorio Privado de la Cañada - Cordoba, Córdoba
  - Sanatorio Privado Duarte Quiroz De Clinica Colombo SA, Córdoba
- Australia (5):
  - Westmead Hospital, Sydney, New South Wales
  - Mater Hospital Brisbane, South Brisbane, Queensland
  - Gold Coast University Hospital, Southport, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Royal Melbourne Hospital, Parkville, Victoria
- Austria (4):
  - Kepler Universitatsklinikum Med Campus III, Linz
  - KH der Barmherzigen Brüder Linz, Linz
  - Medizinische Universitaet Wien, Medizinische Klinik I, Abteilung für Infektionskrankheiten und Tropenmedizin, Vienna
  - Klinik Favoriten (Sozialmedizinisches Zentrum Sued - Kaiser-Franz-Josef-Spital mit Gottfried von Preyer'schem Kinderspital), Vienna
- Germany (5):
  - Albeilung für Kardiologie und Pneumologie, Dachau, Bavaria
  - Medizinische Hochschule, Hanover, Lower Saxony
  - Universitaetsklinikum Carl Gustav Carus TU Dresden, Dresden, Saxony
  - Universitätsmedizin Göttingen, Göttingen, Südniedersachsen
  - Universitaetsklinikum Jena, Jena, Thuringia
- Italy (20):
  - UOC Malattie dell'Apparato Respiratorio, Policlinico di Bari, Bari
  - ASST - Ospedale Papa Giovanni XXIII - UOC Pneumologia, Bergamo
  - Azienda Ospedaliera Universitaria di Bologna - Ospedale Sant'Orsola, Bologna
  - Campus Universitario "Salvatore Venuta", Complesso Clinico, Padiglione B, 8° livello, Pneumologia, Catanzaro
  - Azienda Ospedaliera Universitaria Arcispedale Sant'Anna, Ferrara
  - University Of Genoa - Ospedale Policlinico IRCCS San Martino di Genova, Genova
  - IRCCS Istituto Clinico Humanitas U.O. Medicina D'Urgenza, Milan
  - IRCCS Ospedale San Raffaele Centro di Ricerca Anestesia e Rianimazione, Milan
  - ASST SANTI PAOLO E CARLO Ospedale San Paolo Struttura Complessa Malattie Infettive, Milan
  - Università degli Studi di Milano-Ospedale "L.Sacco" Polo Universitario - ASST Fatebenefratelli Sacco, Milan
  - ASST Grande Ospedale Metropolitano Niguarda Dipartimento Malattie Infettive, Milan
  - Fondazione Ca' Granda Policlinico Milano, Milan
  - ASST-Monza Ospedale San Gerardo Malattie Infettive, Monza
  - Azienda Ospedaliera Universitaria Federico II., Napoli
  - Clinica Pneumologica "L. Vanvitelli" - Osp Monaldi, Napoli
  - Università degli Studi della Campania "Luigi Vanvitelli", Napoli
  - Università degli studi di Padova, Unità Malattie Respiratorie, Padua
  - AOUP "P.Giaccone" - UOC Pneumologia, Palermo
  - Fondazione IRCCS Policlinico San Matteo - UOC Pneumologia, Dipartimento di Scienze Mediche e Malattie Infettive, Pavia
  - Struttura semplice di terapia demi-intensiva respiratoria S.C. di pneumologia AO IRCCS Santa Maria Nuova, Reggio Emilia
- Turkey (Türkiye) (9):
  - Ankara City Hospital, Ankara
  - Dicle University, Medical Faculty, Diyarbakır
  - Gaziantep Universitesi Sahinbey Arastirma Ve Uygulama Hastanesi, Gaziantep
  - Acibadem Atakent Hospital, Istanbul
  - Dokuz Eylul University Faculty of Medicine, Izmir
  - Kayseri State Hospital, Kayseri
  - Kocaeli Universitesi Tip Fakultesi, Kocaeli
  - Inonu Uni.Med.Faculty, Malatya
  - Karadeniz Tecnical Uni. Med. Fac., Trabzon

REFERENCES:
- [Derived] Truwit JD, Fleming K, Nanchal RS. Empowering Respiratory Therapists to Restrict Nebulized 3% Saline and N-Acetylcysteine During Mechanical Ventilation. Respir Care. 2025 Aug;70(8):937-945. doi: 10.1089/respcare.12586. Epub 2025 Feb 24. PMID 40028879